CLINICAL TRIAL: NCT05815108
Title: Prevalence and Prognostic Value of Epstein Barr Virus (EBV) Infection in Patients With Radiologically Isolated Syndrome (RIS)
Brief Title: Epstein Barr Virus Infection in Patients With Radiologically Isolated Syndrome
Acronym: EBV-RIS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23Neuro01
Record Dates: First submitted 2023-03-08; First posted 2023-04-18 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis; Radiologically Isolated Syndrome; Epstein-Barr Virus
MeSH Terms: conditions — Multiple Sclerosis; Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RIS Patient: RIS patients validated by the RIS expert group
  Interventions: Other: NO INTERVENTION

INTERVENTIONS:
Other: NO INTERVENTION — NO INTERVENTION

SUMMARY:
The clinical course of RRMS patients is variable. Among RIS-Consortium international cohorts, one third of RIS patients progressed to MS at 5 years and 52.2% at 10 years. Biomarkers predictive of MS conversion are key elements to organize personalized medical care, for both follow-up and treatment strategies. EBV seems to be an interesting candidate regarding its involvement MS pathophysiology. It can be easily assess in blood sample in contrast to others prognostic biomarkers validated in RIS : oligoclonal bands and NfL levels in cerebrospinal fluid and serum. In RIS, treatment targeting EBV could significantly modify the course of the disease. The investigators aim to make the fisrt description of the EBV epidemiology (immunoglobulin (Ig)M and IgG anti-viral capsid antigen (VCA), IgG anti Epstein-Barr nuclear antigen (EBNA)) among RIS patients and to investigate a correlation between the different antibodies' titers (IgM VCA, IgG VCA, IgG EBNA) and the course of the disease (clinical conversion or evidence of disease activity (EDA)).

ELIGIBILITY:
Inclusion Criteria:

Patients with RIS confirmed by the RIS expert center of the Nice CHU; EBNA status at RIS diagnosis available

Exclusion Criteria:

none

Ages: 15 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with RIS confirmed by the RIS expert center of the Nice CHU, included in the international cohort of the RIS Consortium for which retrospective serological data are available.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Comparaison of IgG EBNA status at RIS diagnostic in patients who remain RIS and those who develop MS according to their conversion delay | Retrospectively at baseline (RIS diagnosis)
  IgG EBNA (negative/positive)

SECONDARY OUTCOMES:
Comparaison of IgM VCA EBNA status at RIS diagnostic in patients who remain RIS and those who develop MS according to their conversion delay | Retrospectively at baseline (RIS diagnosis) and through study completion, an average of 5 years.
  quantity of IgM VCA EBNA (U/ml)
Comparaison of IgG VCA EBNA status at RIS diagnostic in patients who remain RIS and those who develop MS according to their conversion delay | Retrospectively at baseline (RIS diagnosis) and through study completion, an average of 5 years.
  quantity of IgM VCA EBNA (U/ml)
Prevalence of EBV seropositivity in RIS patients according to their MRI activity | Retrospectively at baseline (RIS diagnosis) and through study completion, an average of 5 years.
  EBV seropositivity (negative/positive) according clinical event and Dissemination in time and in space
Prevalence of EBV seropositivity in RIS patients according to their clinical and/or MRI activity (EDA) | Retrospectively at baseline (RIS diagnosis) and through study completion, an average of 5 years.
  EBV seropositivity (negative/positive) according clinical event and Dissemination in time and in space
Assessment correlation between antibodies titers and clinical conversion | Retrospectively at baseline (RIS diagnosis) and through study completion, an average of 5 years.
  quantity of IgG VCA EBNA (U/ml) and IgM VCA EBNA (U/ml) according Dissemination in time and in space
Assessment correlation between antibodies titers and clinical and/or MRI activity (EDA) | Retrospectively at baseline (RIS diagnosis) and through study completion, an average of 5 years.
  quantity of IgG VCA EBNA (U/ml) and quantity of IgM VCA EBNA (U/ml) according clinical event and Dissemination in time and in space

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No